CLINICAL TRIAL: NCT05149079
Title: Randomized, Double Blind, Placebo Controlled Clinical Study to Investigate the Effect of a Marine Protein Hydrolysate in Healthy Adults
Brief Title: Effects of a Marine Protein Hydrolysate in Healthy Adults
Acronym: MARPEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Alesund Hospital (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FHF-Study
Record Dates: First submitted 2021-03-09; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Healthy Diet
Keywords: Cardiovascular disease risk; Protein supplementation; Metabolic health

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled clinical study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The groups will be randomly labelled A or B. Neither participants, care providers or statistician will know the treatments of the groups before the statistical analyses for the primary outcome have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (whey protein supplement) (Placebo Comparator): Participants will consume 18 g of the placebo whey protein supplement each day for 12 weeks.
  Interventions: Dietary Supplement: Placebo
- Cod protein hydrolysate supplement (Active Comparator): Participants will consume 18 g of the cod protein supplement each day for 12 weeks.
  Interventions: Dietary Supplement: Cod protein hydrolysate

INTERVENTIONS:
Dietary Supplement: Cod protein hydrolysate — Rest raw materials (RRM) from cod (Fjordlaks AS, Norway) are used for the hydrolysis production (Food Grade). Freshly minced RRM is treated wth enzymes optimized to generate bioactive hydrolysates using facilities and techniques approved for human consumption.
  Arms: Cod protein hydrolysate supplement
Dietary Supplement: Placebo — Whey protein powder, commercially available
  Other Names: Whey protein powder
  Arms: Placebo (whey protein supplement)

SUMMARY:
This randomized, double blind, controlled trial investigates changes in the cardiovascular index (triacylglycerol/HDL-cholesterol × waist/hip ratio) after 12 weeks of marine protein hydrolysate (MPH) or whey protein powder (placebo) supplementation in adult healthy persons. Additionally, the study investigates potential effects on plasma parameters of metabolic health including lipids, glucose, inflammatory parameters and redox state, as well as associations between dietary MPH and body weight, abdominal obesity, body composition, and gut microbiota composition. Finally, putative end-products of diet-microbial interactions (TMAO and short-chain fatty acids) with CVD risk factors and biomarkers of mitochondrial function are examined.

DETAILED DESCRIPTION:
Marine protein sources, including fish and fish protein hydrolysates, may have particular health benefits. Health benefits from fish consumption have been attributed to the n-3 polyunsaturated fatty acids, in particular eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). Proteins from marine sources may contain valuable bioactive components, with amino acid composition and protein profiles that differ from terrestrial sources. Generally, the dietary source of protein can affect cellular energy metabolism, and hydrolyzed peptides can have potent and specific bioactive potential.

Rest raw materials (RRM) from cod (Fjordlaks AS, Norway) are used for the hydrolysis production (Food Grade). Freshly minced RRM were treated with enzymes optimized to generate bioactive hydrolysates using facilities and techniques approved for human consumption. The investigational products are given in a dose of 18 g protein per day, corresponding to the protein content of a standard meal, and similar to doses recommended in a range of protein supplements.

The study enrolls around 70 men and women age of 20-80 years with waist circumference of < 102 cm for men and < 88 cm for women. Prospective study participants were informed of the study and invited to participate through advertising primarily in social media (Facebook advertisement, geographically limited to 12 km surrounding the city centers of Bergen and Ålesund). Participants provided written informed consent, and were screened via self-reporting in an online form in EasyTrial hosted by the Research Unit for Clinical Trials at the University of Bergen. Data collection by the study staff at baseline verifies inclusion and exclusion criteria and participant eligibility prior to randomization. The potential participants are informed about practical details at a digital or physical meeting 1-2 weeks prior to baseline.

Groups of participants (40-60% males/females) are block randomized to the two treatments using randomly selected block sizes, and stratified according to sex.

The participants are given a container with the powder sufficient for the entire study period, and a spoon to measure the intake at breakfast (6 g), lunch (6 g) and supper (6 g), or morning (9 g) and evening (9 g) according to individual preference. The patients will mix the powder products in water or mineral water. Flavours have been masked by supplementation with beet powder, and mixing 0.5 g fish hydrolysate per serving in the placebo, to minimize differences in taste of the placebo and active product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects at age 20-80 years old understanding Norwegian oral and written information
* Waist circumference for males < 102 cm and females < 88 cm

Exclusion Criteria:

* Pregnancy or lactation
* Having used high-dose omega-3 PUFA supplements (>2 g/day) less than 28 days prior to randomization
* Use of corticosteroids that will influence protein metabolism
* Antibiotic treatment previous 3 months
* Alcohol or drug abuse or any conditions associated with poor compliance
* Medical diagnosis of malabsorption disorders, Crohn's disease, or lactose intolerance
* Scheduled hospitalization during the course of the study that could compromise the study
* Diabetes type I or II, serious high blood pressure at screening, serious infections, diseases requiring medication that can influence the study
* Known or suspected sensitivity or allergic reactions to the IMP or excipients
* Presence of other major medical or psychiatric illness that would affect the ability to participate in the study or put the subject at increased risk
* Intake of statins. If needed to obtain the recruitment goals, we will accept people using a low dose of statin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in the cardiovascular index (triacylglycerol/high density lipoprotein (HDL)-cholesterol × waist/hip ratio) | Baseline to 12 weeks
  Triacylclygerol and HDL-cholesterol concentrations will be measured in serum. Waist and hip circumference will be measured using anthropometric tape over light clothing. For waist circumference, the minimum circumference between the iliac crest and the rib cage will be used. For waist circumference the circumference at the level of the greatest protrusion of the buttocks is used.

SECONDARY OUTCOMES:
Changes in the Quick1 index, a surrogate marker of insulin sensitivity | Baseline to 12 weeks
  Measured in serum and calculated as 1 / (log(fasting insulin μU/mL) + log(fasting glucose mg/dL)
Changes in fasting insulin | Baseline to 12 weeks
  Measured in serum
Changes in fasting insulin C-peptide | Baseline to 12 weeks
  Measured in serum
Changes in fasting glucose | Baseline to 12 weeks
  Measured in serum
Changes in total cholesterol | Baseline to 12 weeks
  Measured in serum
Changes in non-high density lipoprotein (HDL) cholesterol | Baseline to 12 weeks
  Measured in serum
Changes in non-esterified fatty acids (NEFA) | Baseline to 12 weeks
  Measured in serum
Changes in triacylglycerol (TAG) | Baseline to 12 weeks
  Measured in serum
Changes in gut microbiota composition | Baseline to 12 weeks
  Measured by 16S sequencing
Changes in short chained fatty acids (SCFA) | Baseline to 12 weeks
  Faecal SCFA concentrations calculated as (mmol/L) × wet faecal weight x faecal moisture content (g/100 g) × 10
Changes in fat mass/fat free mass ratio | Baseline to 12 weeks
  Body composition measured by bioimpedance analysis
Changes in waist-hip ratio | Baseline to 12 weeks
  Waist and hip circumference will be measured using anthropometric tape over light clothing. For waist circumference, the minimum circumference between the iliac crest and the rib cage will be used. For waist circumference the circumference at the level of the greatest protrusion of the buttocks is used
Changes in waist-to-height ratio (WHtR) | Baseline to 12 weeks
  Waist circumference will be measured using anthropometric tape over light clothing. Hight will be measured using a stadiometer. For waist circumference, the minimum circumference between the iliac crest and the rib cage will be used.
Changes in blood pressure | Baseline to 12 weeks
  Blood pressure measurement will be performed manually by a trained nurse using standard equipment
Changes in heart rate | Baseline to 12 weeks
  Heart rate will be determined manually by a trained nurse
Changes in glucagon-like peptide 1 (GLP-1, hormone involved in appetite and metabolism regulation) | Baseline to 12 weeks
  Measured in plasma by ELISA (enzyme-linked immunosorbent assay)
Changes in gastric inhibitory polypeptide (GIP, hormone involved in metabolism regulation) | Baseline to 12 weeks
  Measured in plasma by ELISA (enzyme-linked immunosorbent assay)
Changes in ghrelin (hormone involved in appetite regulation) | Baseline to 12 weeks
  Measured in plasma by ELISA (enzyme-linked immunosorbent assay)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf K Berge, PhD, Study Director — University of Bergen, Norway
Locations (1):
- Research Unit for Health Trials, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SK, Ngo DH, Vo TS. Marine fish-derived bioactive peptides as potential antihypertensive agents. Adv Food Nutr Res. 2012;65:249-60. doi: 10.1016/B978-0-12-416003-3.00016-0. PMID 22361192
- [Background] Erdmann K, Cheung BW, Schroder H. The possible roles of food-derived bioactive peptides in reducing the risk of cardiovascular disease. J Nutr Biochem. 2008 Oct;19(10):643-54. doi: 10.1016/j.jnutbio.2007.11.010. Epub 2008 May 20. PMID 18495464